CLINICAL TRIAL: NCT03718299
Title: An Open-Label, Real World Study Evaluating the Long-Term Quality of Life of Tildrakizumab in Adult Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Real World Study Evaluating the Long-Term Quality of Life of Tildrakizumab in Adult Patients With Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIL2018-1
Record Dates: First submitted 2018-10-15; First posted 2018-10-24 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tildrakizumab 100 mg (Other)
  Interventions: Drug: Injections of tildrakizumab

INTERVENTIONS:
Drug: Injections of tildrakizumab — given at Week 0, Week 4, Week 16, Week 28, Week 40 and Week 52

SUMMARY:
This is a Phase 4 multicenter, uncontrolled open-label study design. There will be a total of 10 study visits at Screening, Baseline, Week 4, Week 8, Week 12, Week 16, Week 28, Week 40, Week 52 and Week 64, with subjects receiving tildrakizumab injections at Week 0, Week 4, Week 16, Week 28, Week 40, and Week 52. The total study duration will be approximately 64 weeks, excluding a screening period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are non-immunocompromised males or females 18 years of age or older.
2. Subjects have ≥3% total body surface area plaque psoriasis.
3. Subjects are candidates for phototherapy or systemic therapy.
4. Subject must be diagnosed at least 6 months prior to entering the study.
5. Females must be surgically sterile, postmenopausal for >5 years, or using a highly effective form of birth control (<1% failure rate), for at least 30 days prior to test article exposure, with a negative serum pregnancy test.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject is younger than 18 years of age.
3. Subjects with uncontrolled mental illness or active suicidal ideations based on baseline mental health questionnaire of choice.
4. Subject is known, or suspected of being unable to comply with the study protocol, in the opinion of the investigator.
5. Subject is currently enrolled in an investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Therapeutics Clinical Research, San Diego, California
  - Site 02, Grandville, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhutani T, Koo J, Heim J, Bhatia N, Mathew J, Ferro T, Vasquez JG. Improvements in Psoriasis-Related Work Productivity with Tildrakizumab: Results from a Phase 4 Real-World Study in Patients with Moderate-to-Severe Plaque Psoriasis. Dermatol Ther (Heidelb). 2024 Apr;14(4):1019-1025. doi: 10.1007/s13555-024-01131-1. Epub 2024 Apr 4. PMID 38575729

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tildrakizumab 100 mg
Started | 55
Completed | 45
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (15.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Quality of Life Measured by Change From Baseline in Psychological General Well-Being Scale
Description: The Psychological General Well-Being scale is a self-administered validated psychometric instrument that measures a person's emotional well-being. It is specifically designed to be suitable for assessing psychological well being in the general medical population as opposed to a psychiatric population. The 22 questions of the PGWB can be further divided into 6 domains: anxiety, depressed mood, positive well being, self-control, general health, and vitality. The PGWB is graded on a Likert scale, which is commonly used in psychometric questionnaires where the answers range from strongly agree to strongly disagree with gradations in between. Total scores range from 0 to 110, with higher scores indicating better psychological well being. This instrument has been validated and used in many countries on large samples of the general population and on various subsets of medical patients.
  The values reported are change in score from baseline.
Time Frame: baseline, week 28 and week 52
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 78 (14)
  Week 28 | 3.7 (12.36)
  Week 52 | 8.0 (14.06)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Week 52; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Improvement in Quality of Life Measured by Change From Baseline in Psychological General Well-Being Scale Over Time
Description: as for outcome 1
Time Frame: baseline, weeks 4, 8, 12, 16, 40, 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 78.1 (14.06)
  Week 4 | 4.2 (10.40)
  Week 8: number analyzed (Participants) | 53
  Week 8 | 4.2 (12.33)
  Week 12: number analyzed (Participants) | 54
  Week 12 | 4.5 (13.56)
  Week 16: number analyzed (Participants) | 54
  Week 16 | 5.3 (13.36)
  Week 40: number analyzed (Participants) | 48
  Week 40 | 5.6 (12.48)
  Week 64: number analyzed (Participants) | 45
  Week 64 | 5.6 (14.14)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p = 0.011, t-test, 2 sided

3. Secondary Outcome: Improvement in Quality of Life Measured by Change From Baseline in Dermatology Life Quality Index Over Time
Description: The DLQI is a self-administered and user-friendly validated questionnaire used to measure the health-related quality of life of adult patients suffering from a skin disease. The items of the DLQI encompass aspects such as symptoms and feelings, daily activities, leisure, work or school, personal relationships and the side effects of treatment.
  Higher scores mean greater impairment of patient's QoL. The DLQI or Dermatology Life Quality Index measures patient's quality of life. The score ranges from 0 to 30. Lower scores indicate less impairment in quality of life
Time Frame: week 64
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 45
score on a scale | -8.0 (5.18)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Proportion of Subjects With Dermatology Life Quality Index Score of 0 or 1
Description: The DLQI is a self-administered and user-friendly validated questionnaire used to measure the health-related quality of life of adult patients suffering from a skin disease. The items of the DLQI encompass aspects such as symptoms and feelings, daily activities, leisure, work or school, personal relationships and the side effects of treatment.
  Higher scores mean greater impairment of patient's QoL. The DLQI or Dermatology Life Quality Index measures patient's quality of life. The score ranges from 0 to 30. Lower scores indicate less impairment in quality of life.
  For 'Units of Measure'- Data entered is percentage of participants, which is calculated by multiplying the value obtained (Proportion in this case) by 100.
Time Frame: baseline, weeks 4, 8, 12, 16, 28, 40, 52, 64
Population: The intent-to-treat (ITT) population
Measure: Number; unit: Percentage of subjects
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
Percentage of subjects
  Baseline | 1.8
  Week 4 | 18.2
  Week 8: number analyzed (Participants) | 52
  Week 8 | 36.5
  Week 12: number analyzed (Participants) | 52
  Week 12 | 42.3
  Week 16: number analyzed (Participants) | 54
  Week 16 | 51.9
  Week 28: number analyzed (Participants) | 53
  Week 28 | 52.8
  Week 40: number analyzed (Participants) | 48
  Week 40 | 58.3
  Week 52: number analyzed (Participants) | 48
  Week 52 | 56.3
  Week 64: number analyzed (Participants) | 45
  Week 64 | 62.2
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; Clopper-Pearson = 62.2, 95% CI 2-sided [46.5 to 76.2]

5. Secondary Outcome: Proportion of Subjects With Dermatology Life Quality Index Score ≤ 5
Description: as for outcome 4
Time Frame: Baseline, weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Number; unit: Percentage of subjects
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
Percentage of subjects
  Baseline | 13
  Week 4 | 56.4
  Week 8: number analyzed (Participants) | 52
  Week 8 | 84.6
  Week 12: number analyzed (Participants) | 52
  Week 12 | 86.5
  Week 16: number analyzed (Participants) | 54
  Week 16 | 88.9
  Week 28: number analyzed (Participants) | 53
  Week 28 | 94.3
  Week 40: number analyzed (Participants) | 48
  Week 40 | 91.7
  Week 52: number analyzed (Participants) | 48
  Week 52 | 89.6
  Week 60: number analyzed (Participants) | 45
  Week 60 | 93.3
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; Clopper-Pearson = 93.3, 95% CI 2-sided [81.7 to 98.6]

6. Secondary Outcome: Proportion of Subjects With a Reduction of ≥ 5 Points in Dermatology Life Quality Index From Baseline
Description: as for outcome 4
Time Frame: baseline, weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Number; unit: Percentage of subjects
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
Percentage of subjects
  Week 4: number analyzed (Participants) | 45
  Week 4 | 44.4
  Week 8: number analyzed (Participants) | 42
  Week 8 | 61.9
  Week 12: number analyzed (Participants) | 42
  Week 12 | 69.0
  Week 16: number analyzed (Participants) | 44
  Week 16 | 75.0
  Week 28: number analyzed (Participants) | 43
  Week 28 | 81.4
  Week 40: number analyzed (Participants) | 40
  Week 40 | 87.5
  Week 52: number analyzed (Participants) | 40
  Week 52 | 82.5
  Week 64: number analyzed (Participants) | 38
  Week 64 | 78.9
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; Clopper-Pearson = 78.9, 95% CI 2-sided [62.7 to 90.4]

7. Secondary Outcome: Changes From Baseline in Percent Affected Body Surface Area
Description: The percent BSA affected with psoriasis will be estimated at each study visit. The investigator may use the estimate that 1% BSA is equivalent to the area of the subject's closed hand (palm with fingers held together).
Time Frame: Weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: Percent BSA
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
Percent BSA
  Baseline | 14.5 (11.54)
  Week 4 | -2.9 (5.70)
  Week 8: number analyzed (Participants) | 50
  Week 8 | -8.7 (11.89)
  Week 12: number analyzed (Participants) | 51
  Week 12 | -10.1 (12.09)
  Week 16: number analyzed (Participants) | 54
  Week 16 | -10.9 (11.57)
  Week 28: number analyzed (Participants) | 52
  Week 28 | -10.9 (12.74)
  Week 40: number analyzed (Participants) | 48
  Week 40 | -11.3 (12.93)
  Week 52: number analyzed (Participants) | 47
  Week 52 | -11.5 (12.79)
  Week 64: number analyzed (Participants) | 45
  Week 64 | -12.7 (11.88)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Static Physician's Global Assessment
Description: The sPGA is used to determine the overall severity of psoriasis lesions at a given time point. Its score ranges from 0 to 5 with higher scores indicating greater severity.
Time Frame: Weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 3.2 (0.56)
  Week 4 | -1.1 (0.71)
  Week 8: number analyzed (Participants) | 50
  Week 8 | -1.8 (0.94)
  Week 12: number analyzed (Participants) | 51
  Week 12 | -2.0 (1.08)
  Week 16: number analyzed (Participants) | 54
  Week 16 | -1.9 (0.80)
  Week 28: number analyzed (Participants) | 52
  Week 28 | -2.0 (1.05)
  Week 40: number analyzed (Participants) | 48
  Week 40 | -2.2 (1.00)
  Week 52: number analyzed (Participants) | 47
  Week 52 | -2.1 (1.07)
  Week 64: number analyzed (Participants) | 45
  Week 64 | -2.2 (1.00)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

9. Secondary Outcome: Changes From Baseline Body Surface Area x Physician's Global Assessment Over Time
Description: The metric of BSA x sPGA is a multiplication of the percentage BSA covered and the sPGA score.
  The scale range for the sPGA is 0 to 5. The scale range for BSA in this study was >=3% (inclusion criterion), which means that it has to be at least 3%, and it can be as high as 100% hypothetically. So the minimum score for sPGA x BSA = 0, and the maximum score is 5 x 100 = 500. So the range for sPGA x BSA in this study was 0 to 500.
  The BSA has a range of 0% to 100% where higher percentages indicate a worse outcome or worse disease
  The sPGA has a range of 0 (clear) to 5 (severe) where higher values indicate a worse outcome or worse disease.
  sPGA is used to determine the overall severity of psoriasis lesions at a given time point. Its score ranges from 0 to 5. BSA covered is reported as percent of body surface area covered. Total score for BSA x sPGA ranges from 0 to 500 with higher scores indicating greater severity.
Time Frame: weeks 4, 8, 12, 16, 28, 40, 52, 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Week 4 | -21.1 (27.47)
  Week 8: number analyzed (Participants) | 50
  Week 8 | -37.1 (42.52)
  Week 12: number analyzed (Participants) | 51
  Week 12 | -38.1 (43.36)
  Week 16: number analyzed (Participants) | 54
  Week 16 | -39.9 (41.74)
  Week 28: number analyzed (Participants) | 52
  Week 28 | -37.8 (45.28)
  Week 40: number analyzed (Participants) | 48
  Week 40 | -38.2 (44.48)
  Week 52: number analyzed (Participants) | 47
  Week 52 | -40.0 (44.33)
  Week 64: number analyzed (Participants) | 45
  Week 64 | -43.3 (41.86)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Changes From Baseline Psoriasis Area Severity Index (% of Psoriasis Area Severity Index Improvement From Baseline, Absolute Psoriasis Area Severity Index ) Over Time
Description: The PASI is a quantitative rating scale for measuring the severity of psoriatic lesions based on area coverage and plaque appearance. PASI analyzes the four regions of the body (head, trunk, upper and lower limbs). It ranges from 0 to 72 with higher scores indicating greater severity.
Time Frame: baseline, weeks 4,16, 28 and 52
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 11.6 (7.12)
  Week 4 | -5.1 (4.60)
  Week 16: number analyzed (Participants) | 54
  Week 16 | -9.3 (7.03)
  Week 28: number analyzed (Participants) | 52
  Week 28 | -9.4 (6.95)
  Week 52: number analyzed (Participants) | 46
  Week 52 | -10.0 (7.32)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Itch-Numeric Rating Scale
Description: The Itch-Numerical Rating Scale (I-NRS) is a simple, 11-point self-administered numeric rating scale. A score of 0 indicates no itch and score of 10 indicates indicates worst imaginable itch
Time Frame: baseline, weeks 4, 8, 12, 16, 28, 40, 52, 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 6.6 (2.57)
  Week 4 | -1.7 (2.47)
  Week 8: number analyzed (Participants) | 53
  Week 8 | -2.8 (3.11)
  Week 12: number analyzed (Participants) | 54
  Week 12 | -3.0 (3.22)
  Week 16: number analyzed (Participants) | 54
  Week 16 | -3.8 (2.84)
  Week 28: number analyzed (Participants) | 53
  Week 28 | -3.8 (3.12)
  Week 40: number analyzed (Participants) | 48
  Week 40 | -3.7 (2.99)
  Week 52: number analyzed (Participants) | 48
  Week 52 | -4.1 (3.06)
  Week 64: number analyzed (Participants) | 45
  Week 64 | -4.4 (2.66)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Scaling-Numeric Rating Scale
Description: The Scaling-NRS (S-NRS) is a simple, 11-point self-administered numeric rating scale that is administered at each visit. A score of 0 represents 'no scaling' and a score of 10, indicates 'worst scaling imaginable'.
Time Frame: Weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 7.0 (2.33)
  Week 4 | -2.6 (2.38)
  Week 8: number analyzed (Participants) | 53
  Week 8 | -4.1 (3.03)
  Week 12: number analyzed (Participants) | 54
  Week 12 | -4.3 (2.95)
  Week 16: number analyzed (Participants) | 54
  Week 16 | -4.5 (2.54)
  Week 28: number analyzed (Participants) | 53
  Week 28 | -4.7 (2.78)
  Week 40: number analyzed (Participants) | 48
  Week 40 | -4.5 (2.86)
  Week 52: number analyzed (Participants) | 48
  Week 52 | -4.6 (2.86)
  Week 64: number analyzed (Participants) | 45
  Week 64 | -4.6 (2.89)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Pain-Numeric Rating Scale
Description: The P-NRS is a simple, 11-point self-administered numeric rating scale. A score of 0 indicates no pain. A score of 10 indicates worst pain imaginable
Time Frame: Weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 3.8 (3.22)
  Week 4 | -1.2 (2.65)
  Week 8: number analyzed (Participants) | 53
  Week 8 | -1.8 (3.18)
  Week 12: number analyzed (Participants) | 54
  Week 12 | -1.8 (2.88)
  Week 16: number analyzed (Participants) | 54
  Week 16 | -2.2 (2.88)
  Week 28: number analyzed (Participants) | 53
  Week 28 | -2.3 (3.05)
  Week 40: number analyzed (Participants) | 48
  Week 40 | -2.3 (2.48)
  Week 52: number analyzed (Participants) | 48
  Week 52 | -2.5 (2.76)
  Week 64: number analyzed (Participants) | 45
  Week 64 | -2.8 (2.75)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

14. Secondary Outcome: Proportion of Patients With Itch Score of 0
Description: The Itch-Numerical Rating Scale (I-NRS) is a simple, 11-point self-administered numeric rating scale. A score of 0 indicates no itch and score of 10 indicates indicates worst imaginable itch.
  For 'Units of Measure'- Data entered is percentage of participants, which is calculated by multiplying the value obtained (Proportion in this case) by 100
Time Frame: weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
Percentage of participants
  Baseline | 1.8
  Week 4 | 3.6
  Week 8: number analyzed (Participants) | 53
  Week 8 | 11.3
  Week 12: number analyzed (Participants) | 54
  Week 12 | 22.2
  Week 16: number analyzed (Participants) | 54
  Week 16 | 16.7
  Week 28: number analyzed (Participants) | 53
  Week 28 | 20.8
  Week 40: number analyzed (Participants) | 48
  Week 40 | 22.9
  Week 52: number analyzed (Participants) | 48
  Week 52 | 22.9
  Week 64: number analyzed (Participants) | 45
  Week 64 | 24.4
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; Mean (Clopper-Pearson) = 24.4, 95% CI 2-sided [12.9 to 39.5]

15. Secondary Outcome: Proportion of Patients With Scaling Score of 0
Description: The Scaling-NRS (S-NRS) is a simple, 11-point self-administered numeric rating scale that is administered at each visit. A score of 0 represents 'no scaling' and a score of 10, indicates 'worst scaling imaginable'.
  For 'Units of Measure'- Data entered is percentage of participants, which is calculated by multiplying the value obtained (Proportion in this case) by 100
Time Frame: Weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
percentage of participants
  Baseline | 0
  Week 4 | 3.6
  Week 8: number analyzed (Participants) | 53
  Week 8 | 20.8
  Week 12: number analyzed (Participants) | 54
  Week 12 | 16.7
  Week 16: number analyzed (Participants) | 54
  Week 16 | 20.4
  Week 28: number analyzed (Participants) | 53
  Week 28 | 22.6
  Week 40: number analyzed (Participants) | 48
  Week 40 | 22.9
  Week 52: number analyzed (Participants) | 48
  Week 52 | 25.0
  Week 64: number analyzed (Participants) | 45
  Week 64 | 17.8
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; Mean (Clopper-Pearson) = 17.8, 95% CI 2-sided [8.0 to 32.1]

16. Secondary Outcome: Proportion of Patients With Pain Score of 0
Description: The P-NRS is a simple, 11-point self-administered numeric rating scale. A score of 0 indicates no pain. A score of 10 indicates worst pain imaginable.
  For 'Units of Measure'- Data entered is percentage of participants, which is calculated by multiplying the value obtained (Proportion in this case) by 100.
Time Frame: Weeks 4, 8, 12, 16, 28, 40, 52, and 64
Population: The intent-to-treat (ITT) population
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
Percentage of participants
  Baseline | 12.7
  Week 4 | 21.8
  Week 8: number analyzed (Participants) | 53
  Week 8 | 34.0
  Week 12: number analyzed (Participants) | 54
  Week 12 | 48.1
  Week 16: number analyzed (Participants) | 54
  Week 16 | 40.7
  Week 28: number analyzed (Participants) | 53
  Week 28 | 50.9
  Week 40: number analyzed (Participants) | 48
  Week 40 | 54.2
  Week 52: number analyzed (Participants) | 48
  Week 52 | 52.1
  Week 64: number analyzed (Participants) | 45
  Week 64 | 48.9
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; Clopper-Pearson = 48.9, 95% CI 2-sided [33.7 to 64.2]

17. Secondary Outcome: Improvement From Baseline in Work Productivity Measured by Change in Work Productivity and Activity Impairment Scale Over Time
Description: The WPAI is a validated, subject-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to general health or a specific health problem. WPAI surveys were analyzed based on published algorithms to determine the following: current employment status, absenteeism, presenteeism, total activity impairment , and total work productivity impairment. Each WPAI score is expressed as impairment percentages (0-100), with higher scores indicating greater impairment (worse outcomes).
Time Frame: baseline, weeks 16, 28, 40, 52, 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline (Total Activity Impairment) | 29.5 (26.56)
  Week 16 (Total Activity Impairment): number analyzed (Participants) | 53
  Week 16 (Total Activity Impairment) | -20.8 (21.47)
  Week 28 (Total Activity Impairment): number analyzed (Participants) | 53
  Week 28 (Total Activity Impairment) | -24.7 (25.47)
  Week 40 (Total Activity Impairment): number analyzed (Participants) | 48
  Week 40 (Total Activity Impairment) | -26.9 (24.33)
  Week 52 (Total Activity Impairment): number analyzed (Participants) | 48
  Week 52 (Total Activity Impairment) | -20.8 (28.57)
  Week 64 Total Activity Impairment): number analyzed (Participants) | 45
  Week 64 Total Activity Impairment) | -27.8 (22.85)
  Baseline (Total Work Productivity Impairment): number analyzed (Participants) | 41
  Baseline (Total Work Productivity Impairment) | 20.9 (22.21)
  Week 16 (Total Work Productivity Impairment): number analyzed (Participants) | 35
  Week 16 (Total Work Productivity Impairment) | -13.7 (21.02)
  Week 28 (Total Work Productivity Impairment): number analyzed (Participants) | 33
  Week 28 (Total Work Productivity Impairment) | -14.5 (20.45)
  Week 40 (Total Work Productivity Impairment): number analyzed (Participants) | 31
  Week 40 (Total Work Productivity Impairment) | 17.1 (19.33)
  Week 52 (Total Work Productivity Impairment): number analyzed (Participants) | 31
  Week 52 (Total Work Productivity Impairment) | -16.4 (22.42)
  Week 64 (Total Work Productivity Impairment): number analyzed (Participants) | 31
  Week 64 (Total Work Productivity Impairment) | -19.4 (20.81)
  Baseline (Absenteeism): number analyzed (Participants) | 41
  Baseline (Absenteeism) | 1.1 (5.66)
  Week 16 (Absenteeism): number analyzed (Participants) | 35
  Week 16 (Absenteeism) | 0.5 (3.85)
  Week 28 (Absenteeism): number analyzed (Participants) | 33
  Week 28 (Absenteeism) | -0.3 (1.93)
  Week 40 (Absenteeism): number analyzed (Participants) | 31
  Week 40 (Absenteeism) | -0.4 (2.00)
  Week 52 (Absenteeism): number analyzed (Participants) | 31
  Week 52 (Absenteeism) | -0.4 (2.00)
  Week 64 (Absenteeism): number analyzed (Participants) | 31
  Week 64 (Absenteeism) | 0.0 (0.00)
  Baseline (Presenteeism): number analyzed (Participants) | 41
  Baseline (Presenteeism) | 20.5 (21.67)
  Week 16 (Presenteeism): number analyzed (Participants) | 35
  Week 16 (Presenteeism) | -14.0 (20.47)
  Week 28 (Presenteeism): number analyzed (Participants) | 33
  Week 28 (Presenteeism) | -14.2 (20.31)
  Week 40 (Presenteeism): number analyzed (Participants) | 31
  Week 40 (Presenteeism) | -16.8 (19.22)
  Week 52 (Presenteeism): number analyzed (Participants) | 31
  Week 52 (Presenteeism) | -16.1 (22.31)
  Week 64 (Presenteeism): number analyzed (Participants) | 31
  Week 64 (Presenteeism) | -19.4 (20.81)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Total Activity Impairment; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg; Total Work Productivity Impairment; Test type: Superiority; p < 0.001, t-test, 2 sided

18. Secondary Outcome: Assessment of Patient Satisfaction With Treatment Measured by Change From Baseline in Treatment Satisfaction Questionnaire for Medication Over Time
Description: The TSQM is a general measure of treatment satisfaction with medication, suitable for use across a wide variety of medication types and illness conditions. The 14-item TSQM Version 1.4 is a reliable and valid instrument to assess patients' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction. The TSQM domain scores range from 0-100 with higher scores representing higher satisfaction on that domain
Time Frame: baseline, weeks 4, 8, 12, 16, 28, 40, 52, 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Week 4 (Effectiveness) | 59.5 (17.03)
  Week 8 (Effectiveness) | 70.8 (23.12)
  Week 12 (Effectiveness) | 71.0 (22.65)
  Week 16 (Effectiveness) | 73.9 (17.39)
  Week 28 (Effectiveness) | 76.5 (19.93)
  Week 40 (Effectiveness) | 78.4 (16.01)
  Week 52 (Effectiveness) | 78.7 (16.89)
  Week 64 (Effectiveness) | 79.5 (20.06)
  Week 4 (Convenience) | 83.3 (15.89)
  Week 8 (Convenience) | 85.1 (14.33)
  Week 12 (Convenience) | 86.9 (13.70)
  Week 16 (Convenience) | 84.0 (12.57)
  Week 28 (Convenience) | 85.1 (13.42)
  Week 40 (Convenience) | 85.6 (13.93)
  Week 52 (Convenience) | 85.2 (13.58)
  Week 64 (Convenience) | 82.2 (16.35)
  Week 4 (Global Satisfaction) | 72.7 (18.55)
  Week 8 (Global Satisfaction): number analyzed (Participants) | 52
  Week 8 (Global Satisfaction) | 77.5 (21.19)
  Week 12 (Global Satisfaction): number analyzed (Participants) | 54
  Week 12 (Global Satisfaction) | 77.4 (20.89)
  Week 16 (Global Satisfaction): number analyzed (Participants) | 54
  Week 16 (Global Satisfaction) | 79.4 (16.69)
  Week 28 (Global Satisfaction): number analyzed (Participants) | 53
  Week 28 (Global Satisfaction) | 80.5 (17.78)
  Week 40 (Global Satisfaction): number analyzed (Participants) | 48
  Week 40 (Global Satisfaction) | 81.4 (15.15)
  Week 52 (Global Satisfaction): number analyzed (Participants) | 48
  Week 52 (Global Satisfaction) | 81.7 (18.40)
  Week 64 (Global Satisfaction): number analyzed (Participants) | 45
  Week 64 (Global Satisfaction) | 81.9 (20.47)
  Week 4 (Side Effects) | 70.8 (14.61)
  Week 8 (Side Effects) | 78.1 (18.75)
  Week 12 (Side Effects) | 73.4 (11.83)
  Week 16 (Side Effects) | 68.8 (6.25)
  Week 28 (Side Effects) | 81.3 (10.83)
  Week 40 (Side Effects) | 81.3 (6.25)
  Week 52 (Side Effects) | 77.1 (9.55)
  Week 64 (Side Effects) | 79.2 (3.61)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Treatment Satisfaction Questionnaire for Medication over time- Effectiveness; Test type: Superiority; Mean = 79.5, Standard Deviation 20.06
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg; Treatment Satisfaction Questionnaire for Medication over time-Side Effects; Test type: Superiority; p < 0.001, Exact binomial test
Statistical Analysis 3: Comparison: Tildrakizumab 100 mg; Treatment Satisfaction Questionnaire for Medication over time - Convenience; Test type: Superiority; Mean = 82.2, Standard Deviation 16.35
Statistical Analysis 4: Comparison: Tildrakizumab 100 mg; Treatment Satisfaction Questionnaire for Medication over time - Global Satisfaction; Test type: Superiority; Mean = 81.9, Standard Deviation 20.47

19. Secondary Outcome: Assessment of Tildrakizumab Overall Satisfaction Over Time Using Numerical Rating Scales
Description: The Tildrakizumab Overall Satisfaction Scale is an 11-point simple, self-administered numeric rating scale. Subjects indicate their overall satisfaction by circling the integer that best describes their experience on a scale. A score of 0 indicates 'not satisfied' and 10 indicates 'extremely satisfied'.
Time Frame: weeks 4, 8, 12, 16, 28, 40, 52, 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Week 4 (Improvement in Symptoms) | 6.0 (2.36)
  Week 8 (Improvement in Symptoms): number analyzed (Participants) | 53
  Week 8 (Improvement in Symptoms) | 7.6 (2.44)
  Week 12 (Improvement in Symptoms): number analyzed (Participants) | 54
  Week 12 (Improvement in Symptoms) | 7.7 (2.45)
  Week 16 (Improvement in Symptoms): number analyzed (Participants) | 54
  Week 16 (Improvement in Symptoms) | 8.0 (2.03)
  Week 28 (Improvement in Symptoms): number analyzed (Participants) | 53
  Week 28 (Improvement in Symptoms) | 8.0 (2.30)
  Week 40 (Improvement in Symptoms): number analyzed (Participants) | 48
  Week 40 (Improvement in Symptoms) | 8.4 (1.85)
  Week 52 (Improvement in Symptoms): number analyzed (Participants) | 48
  Week 52 (Improvement in Symptoms) | 8.4 (2.15)
  Week 64 (Improvement in Symptoms): number analyzed (Participants) | 45
  Week 64 (Improvement in Symptoms) | 8.7 (2.01)
  Week 4 (Speed of Symptom Improvement) | 5.9 (2.39)
  Week 8 (Speed of Symptom Improvement): number analyzed (Participants) | 53
  Week 8 (Speed of Symptom Improvement) | 7.5 (2.55)
  Week 12 (Speed of Symptom Improvement): number analyzed (Participants) | 54
  Week 12 (Speed of Symptom Improvement) | 7.2 (2.80)
  Week 16 (Speed of Symptom Improvement): number analyzed (Participants) | 54
  Week 16 (Speed of Symptom Improvement) | 7.7 (2.15)
  Week 28 (Speed of Symptom Improvement): number analyzed (Participants) | 53
  Week 28 (Speed of Symptom Improvement) | 7.8 (2.44)
  Week 40 (Speed of Symptom Improvement): number analyzed (Participants) | 48
  Week 40 (Speed of Symptom Improvement) | 8.4 (1.75)
  Week 52 (Speed of Symptom Improvement): number analyzed (Participants) | 48
  Week 52 (Speed of Symptom Improvement) | 7.9 (2.36)
  Week 64 (Speed of Symptom Improvement): number analyzed (Participants) | 45
  Week 64 (Speed of Symptom Improvement) | 8.3 (2.30)
  Week 4 (Frequency of Taking Medication) | 7.8 (2.05)
  Week 8 (Frequency of Taking Medication): number analyzed (Participants) | 53
  Week 8 (Frequency of Taking Medication) | 8.4 (1.75)
  Week 12 (Frequency of Taking Medication): number analyzed (Participants) | 54
  Week 12 (Frequency of Taking Medication) | 8.2 (2.08)
  Week 16 (Frequency of Taking Medication): number analyzed (Participants) | 54
  Week 16 (Frequency of Taking Medication) | 8.2 (2.19)
  Week 28 (Frequency of Taking Medication): number analyzed (Participants) | 53
  Week 28 (Frequency of Taking Medication) | 8.3 (2.24)
  Week 40 (Frequency of Taking Medication): number analyzed (Participants) | 48
  Week 40 (Frequency of Taking Medication) | 8.8 (2.12)
  Week 52 (Frequency of Taking Medication): number analyzed (Participants) | 48
  Week 52 (Frequency of Taking Medication) | 8.8 (2.12)
  Week 64 (Frequency of Taking Medication): number analyzed (Participants) | 45
  Week 64 (Frequency of Taking Medication) | 9.1 (1.70)
  Week 4 (Side Effects) | 8.6 (2.14)
  Week 8 (Side Effects): number analyzed (Participants) | 53
  Week 8 (Side Effects) | 9.0 (1.50)
  Week 12 (Side Effects): number analyzed (Participants) | 54
  Week 12 (Side Effects) | 9.2 (1.48)
  Week 16 (Side Effects): number analyzed (Participants) | 54
  Week 16 (Side Effects) | 9.2 (1.52)
  Week 28 (Side Effects): number analyzed (Participants) | 53
  Week 28 (Side Effects) | 9.1 (1.54)
  Week 40 (Side Effects): number analyzed (Participants) | 48
  Week 40 (Side Effects) | 9.3 (1.59)
  Week 52 (Side Effects): number analyzed (Participants) | 48
  Week 52 (Side Effects) | 9.5 (1.22)
  Week 64 (Side Effects): number analyzed (Participants) | 45
  Week 64 (Side Effects) | 9.6 (0.68)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Improvement in Symptoms; Test type: Superiority; Mean = 8.7, Standard Deviation 2.01
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg; Speed of Symptom Improvement; Test type: Superiority; Mean = 8.3, Standard Deviation 2.30
Statistical Analysis 3: Comparison: Tildrakizumab 100 mg; Frequency of Taking Medication; Test type: Superiority; Mean = 9.1, Standard Deviation 1.70
Statistical Analysis 4: Comparison: Tildrakizumab 100 mg; Side Effects; Test type: Superiority; Mean = 9.6, Standard Deviation 0.68

20. Secondary Outcome: Assessment of Patient Happiness With Psoriasis Control Over Time Using Numerical Rating Scale
Description: The Patient Happiness with Psoriasis Control assessment is an 11-point simple, self- administered numeric rating scale ranging in score from 0 to 10 that is administered at each visit.
  Subjects indicate their overall happiness with psoriasis control by circling the integer that best describes their experience on a scale. A score of 0 indicates 'extremely unhappy'. A score of 10 indicates 'extremely happy'.
Time Frame: weeks 4, 8, 12, 16, 28, 40, 52, 64
Population: The intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tildrakizumab 100 mg
Number analyzed (Participants) | 55
score on a scale
  Baseline | 2.7 (2.33)
  Week 4 | 3.7 (3.65)
  Week 8: number analyzed (Participants) | 53
  Week 8 | 5.1 (3.69)
  Week 12: number analyzed (Participants) | 54
  Week 12 | 5.1 (3.73)
  Week 16: number analyzed (Participants) | 54
  Week 16 | 5.5 (3.41)
  Week 28: number analyzed (Participants) | 53
  Week 28 | 5.7 (2.91)
  Week 40: number analyzed (Participants) | 48
  Week 40 | 5.9 (3.00)
  Week 52: number analyzed (Participants) | 48
  Week 52 | 6.0 (2.78)
  Week 64: number analyzed (Participants) | 45
  Week 64 | 6.0 (2.97)
Statistical Analysis 1: Comparison: Tildrakizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

21. Other Pre Specified Outcome: Treatment-emergent AEs
Description: The reported values are entered in the 'Other Adverse events' section
Time Frame: baseline, weeks 4, 8, 12, 16, 28, 40, 52,,64
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Week 64
Arm/Group | Tildrakizumab 100 mg
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 4/55
Other Adverse Events (participants affected / at risk) | 29/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tildrakizumab 100 mg (N=55)
COVID-19 pneumonia (Infections and infestations) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ischaemic stroke (Nervous system disorders) | 1
IgA nephropathy (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tildrakizumab 100 mg (N=55)
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Large intestine polyp (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Haematuria (Renal and urinary disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03718299/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03718299/SAP_001.pdf